CLINICAL TRIAL: NCT06794463
Title: Turkish Version of Computer Usage Proficiency Questionnaire, Validity and Reliability Study
Brief Title: Turkish Version of Computer Usage Proficiency Questionnaire
Status: Completed | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Principal Investigator, Uludag University
Other Study IDs: 2025/1-5
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-04

CONDITIONS: Geriatric; Technology
Keywords: CPQ; Reliability; Validity; CPQ-TR

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Computer Proficiency Questionnaire (CPQ) assesses older individuals' computer and information technology skills. The questionnaire promotes digital inclusion by tailoring training packages to meet individual requirements. The CPQ serves as a continuous evaluation tool to track participants' progress in digital inclusion initiatives throughout time. The CPQ identifies unique problems that older persons have while utilizing digital technology, allowing for tailored solutions to overcome these barriers.

DETAILED DESCRIPTION:
The adaptation of the elderly population to technology has increased rapidly with demographic changes and developments in the field of Gerontechnology, which supports successful aging by integrating technology into the daily lives of older individuals. Gerontechnology focuses on the development and application of communication and information technologies in order to increase the independence and social participation of older individuals.

Digital competence requires cognitive and technical skills that include processes such as finding, understanding, evaluating, creating and communicating digital information; it is of fundamental importance for the digital society. The Computer Use Competence Survey stands out as an assessment tool that measures the competence of older individuals in using computers and information technologies. This survey supports digital inclusion by contributing to the development of training programs tailored to individual needs. In addition, the Computer Use Competence Survey can be used as a continuous assessment tool to measure the progress of individuals participating in digital inclusion programs over time. Another strength of the Computer Use Competence Survey is that it can identify specific barriers that older individuals encounter when using digital technology and allows for special measures to be taken to overcome these barriers.

The aim of this study is to provide a reliable tool for assessing the digital competence of the elderly population in Turkey by performing the cross-cultural adaptation and content validation of the Computer Use Proficiency Questionnaire in Turkish.

ELIGIBILITY:
Inclusion Criteria:

* Being a native Turkish speaker,
* Having no reading and writing problems,
* Having a desktop or laptop computer,
* Agreeing to participate in the study

Exclusion Criteria:

-Individuals with neurological diseases such as cognitive impairment, Alzheimer's, dementia, etc. will be excluded from the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Geriatric individuals between the ages of 65-80 who can use computers.
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Age of the patients | 1 week
  Age will be recorded.
Gender of the patients | 1 week
  Gender will be recorded.
Computer Usage Proficiency Questionnaire | 1 week
  Computer Usage Proficiency Questionnaire will be filled out under the supervision of a physiotherapist
System Usability Scale | 1 week
  System Usability Scalewill be filled out under the supervision of a physiotherapist

CONTACTS AND LOCATIONS:
Overall Officials: Selim Mahmut GÜNAY, Dr, Study Chair — Uludağ University
Locations (1):
- Uludag University, Bursa, nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided